CLINICAL TRIAL: NCT02294617
Title: Comparative Evaluation of the Perceptions and Utilization of Nicotine Inhalation Devices
Brief Title: E-cigarette vs. Nicotine Inhaler Comparisons
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Michael B. Steinberg, MD, MPH, FACP, Associate Professor of Medicine, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: P30CA072720 (NIH)
Record Dates: First submitted 2014-06-23; First posted 2014-11-19 (Estimated); Last update posted 2025-04-13 (Actual); Status verified 2014-11

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking | interventions — Electronic Nicotine Delivery Systems; Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nicotrol Inhaler (Active Comparator): Subjects will use the Nicotine Inhaler for 3 days.
  Interventions: Other: Nicotrol Inhaler
- Electronic Cigarette (Active Comparator): Subject will use the electronic cigarette for 3 days.
  Interventions: Other: Electronic Cigarette

INTERVENTIONS:
Other: Electronic Cigarette — Subject will use electronic cigarette for 3 days.
  Arms: Electronic Cigarette
Other: Nicotrol Inhaler — Subjects will use the Nicotrol Inhaler for 3 days.
  Arms: Nicotrol Inhaler

SUMMARY:
The goal of this study is to get information from current smokers about how they feel towards both the electronic cigarette (e-cigarette) and the nicotine oral inhaler. This will include beliefs, harms, appeal, ease of use, enjoyment, and their use for helping people stop smoking.

DETAILED DESCRIPTION:
Subjects will be seen at Baseline, then 3-days post-baseline, then 9 days post-baseline for post product use questionnaires and carbon monoxide monitoring. The time frame for follow up is 6 months post Baseline visit.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be smokers 18 years or older, who have had no previous experience with either the e-cigarette or the nicotine oral inhaler, and will be recruited from the local community. They can currently smoke any amount or frequency and with any level of motivation to stop smoking.

Exclusion Criteria:

* Exclusion criteria include recent (within 2 weeks) myocardial infarction or angina, poorly controlled asthma/chronic obstructive pulmonary disease , active substance abuse, pregnancy, or current use of any other cessation medications

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-08; Primary Completion 2014-04 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Satisfaction of devices on Likert Scale | 6 months (August 2012-December 2013)
  The goal of this study is to gather data from current smokers regarding their perceptions and experiences with both the e-cigarette and the nicotine oral inhaler over a 6 month time period.